CLINICAL TRIAL: NCT02069574
Title: Identification of Novel Periodontal Disease Biomarkers Using microRNA Expression in Saliva
Brief Title: Diagnosis of Periodontal Disease Using Genetic Marker in Saliva
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Su-Hwan Kim, Assistant Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013-0940
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- severe periodontitis group (Experimental): non-surgical periodontal therapy
  Interventions: Procedure: non-surgical periodontal therapy
- Moderate periodontitis group (Experimental): non-surgical periodontal therapy
  Interventions: Procedure: non-surgical periodontal therapy
- healthy control (No Intervention): No treatment

INTERVENTIONS:
Procedure: non-surgical periodontal therapy
  Arms: Moderate periodontitis group; severe periodontitis group

SUMMARY:
The purpose of the present study is to identify the novel periodontal disease biomarkers using differentially expressed microRNA in the saliva. The severity of chronic periodontal diseases and the time of pre- and post-treatment are major classification criteria. The obtained data will secure the foundation for the development of a new non-invasive diagnostic methods for early diagnosis & prognosis prediction of periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

A. Severe Periodontal Disease

* Patients with chronic severe periodontitis
* Primary treatment of periodontal scaling, subgingival curettage is required, and the general progress of the protocol agreed with the basic periodontal therapy patients.
* subjects agreed collecting saliva and gingival crevicular fluid and physicochemical tests and genetic testing

A. Moderate Periodontal Disease

* Patients with chronic moderate periodontitis
* Primary treatment of periodontal scaling, subgingival curettage is required, and the general progress of the protocol agreed with the basic periodontal therapy patients.
* subjects agreed collecting saliva and gingival crevicular fluid and physicochemical tests and genetic testing

C. Healthy Control

* Healthy periodontal patients ( more than 20 permanent teeth are present , in all parts of deep periodontal pockets measuring 4mm or less, and height is 2mm or less clinical attachment person)
* subjects agreed collecting saliva and gingival crevicular fluid and physicochemical tests and genetic testing

Exclusion Criteria:

* Received periodontal treatment within the last six months
* recently taken antibiotics within 3 months if you need a prescription antibiotic prophylaxis
* taking the drug can affect periodontal status for a long period of time
* pregnant or breastfeeding
* In case of oral inflammatory mucosal disease (Lichen planus, etc.)
* A history of alcoholism or drug abuse if
* other special systemic disease (high blood pressure)
* ages under 18

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Expression level of MicroRNAs using Microarray | Change from Baseline in expression level of MicroRNAs at 1,6,12 months

SECONDARY OUTCOMES:
Expression level of cytokines using multiple cytokine analysis | Change from Baseline in expression level of cytokines at 1,6,12 months
  * Pro-inflammatory biomarker : interleukin(IL)-1a, IL-1b, IL-6, IL-8
  * Matrix metalloproteinase(MMP) : MMP-8, MMP-9
  * Anti-inflammatory biomarker: IL-10, inhibitor of MMP (TIMP)-1

CONTACTS AND LOCATIONS:
Overall Officials: Su-Hwan Kim, PhD., Principal Investigator — Asan Medical Center
Locations (1):
- ASAN Medical Center, Seoul, South Korea